CLINICAL TRIAL: NCT01390168
Title: Tailored Internet-administrated Treatment of Anxiety Disorders - A Randomised Controlled Trial (NOVA II)
Brief Title: Internet-administrated Treatment of Anxiety Disorders
Acronym: NOVA II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC-FAS-2008-1145
Record Dates: First submitted 2011-07-01; First posted 2011-07-08 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Waiting Lists

ARMS (2):
- tailored internet-administrated CBT (Experimental): Behavioral: tailored internet-administrated CBT
  Interventions: Behavioral: Tailored Internet-administrated CBT-Treatment
- waitlist (Active Comparator): waitlist
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Tailored Internet-administrated CBT-Treatment — This intervention contains up to 6-10 text-based self-help modules in which 4 modules are fixed (the first three and the last) and the rest are "prescribed following the diagnostic telephone interview. These modules contain material on panic disorder, social phobia, stress management, assertiveness training, concentration, relaxation among other things.
  Arms: tailored internet-administrated CBT
Behavioral: Waitlist — active waitlist
  Arms: waitlist

SUMMARY:
The purpose of this study is to determine whether tailored internet-administered cbt is a feasible treatment for anxiety disorders in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* fulfill the criteria for at least one anxiety syndrome

Exclusion Criteria:

* ongoing psychological treatment
* suicidal prone
* ongoing alcohol addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinical Outcome in Routine Evaluation - Outcome Measure (CORE-OM) | Two weeks pre treatment (baseline), two weeks post treatment, and 12 months post treatment
  Measures anxiety and depressive symptoms.
  Change from baseline in anxiety and depressive symptoms expected between time frames.

SECONDARY OUTCOMES:
Change from baseline in Beck Anxiety Inventory (BAI) | Two weeks pre treatment (baseline), two weeks post treatment, 12 months post treatment
  Measures anxiety symtoms.
  Change from baseline in anxiety symptoms expected between time frames.
Change from baseline in Montgomery Åsberg Depression Rating Scale-Self Rated (MADRS-S) | Two weeks pre treatment (baseline), two weeks post treatment, and 12 months post treatment
  Measures depressive symptoms.
  Change from baseline in depressive symptoms expected between time frames.
Change from baseline in Quality of Life Inventory (QOLI) | Two weeks pre treatment (baseline), two weeks post treatment, and 12 months post treatment
  Measures quality of life.
  Change from baseline in quality of life expected between time frames.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Study Director — Umeå University; Gerhard Andersson, Professor, Study Chair — Linkoeping University; Lise Bergman Nordgren, Ph D Student, Study Chair — Linkoeping University
Locations (1):
- Department of Behavioural Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Nordgren LB, Hedman E, Etienne J, Bodin J, Kadowaki A, Eriksson S, Lindkvist E, Andersson G, Carlbring P. Effectiveness and cost-effectiveness of individually tailored Internet-delivered cognitive behavior therapy for anxiety disorders in a primary care population: a randomized controlled trial. Behav Res Ther. 2014 Aug;59:1-11. doi: 10.1016/j.brat.2014.05.007. Epub 2014 Jun 2. PMID 24933451
- [Derived] Nordgren LB, Andersson G, Kadowaki A, Carlbring P. Tailored internet-administered treatment of anxiety disorders for primary care patients: study protocol for a randomised controlled trial. Trials. 2012 Feb 9;13:16. doi: 10.1186/1745-6215-13-16. PMID 22321916